CLINICAL TRIAL: NCT01117922
Title: Philadelphia Collaborative Preterm Prevention Project
Brief Title: Philadelphia Preterm Prevention Project
Acronym: PPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#09-007191
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2010-05

CONDITIONS: Preterm Birth
Keywords: preterm birth; interconceptional intervention; pregnancy outcomes
MeSH Terms: conditions — Premature Birth | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): After consent, subjects will be assigned to either a usual care group (no intervention) or an intervention group (targeted interconceptional interventions).
  Interventions: Other: Psychological intervention
- Usual Care Group (Other): This group will receive usual care.
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Other: Psychological intervention — Subjects will be randomized into either usual care or interconceptional intervention groups. If the subject is randomized into the intervention group, she will receive targeted interventions to reduce one of several risk factors: smoking, depression, infectious disease burden and maternal stress, and achieving an appropriate BMI. A woman who is randomized to the intervention group may receive interventions on one, two, three, four, or five of the targeted intervention methods, depending on her needs.
  Arms: Intervention
Other: Usual Care Group
  Arms: Usual Care Group

SUMMARY:
This is a randomized clinical trial in which all Philadelphia resident women experiencing a pre-term birth (PTB) at <34 weeks of gestation (GA) over an 18 month period will be approached at the time of the postpartum hospital stay. Consenting women will be randomized into a usual care group or an interconceptional intervention targeting five risk conditions, all of which increase systemic inflammation. Our primary objective in this study is to assess the efficacy of our interconceptional intervention on the rate of repeat PTB.

DETAILED DESCRIPTION:
This is a randomized clinical trial in which all Philadelphia resident women experiencing a pre-term birth (PTB) at <34 weeks of gestation (GA) over an 18 month period will be approached at the time of the postpartum hospital stay. Consenting women will be randomized into a usual care group or an interconceptional intervention targeting five risk conditions, all of which increase systemic inflammation. Our primary objective in this study is to assess the efficacy of our interconceptional intervention on the rate of repeat PTB.

Participants will be randomized into one of two groups: usual care of interconceptional intervention. Those who are randomized into the interconceptional intervention group will be targeted for five risk conditions, including smoking, depression, infectious disease burden and maternal stress, and achieving an appropriate BMI. It is hoped that by reducing these seemingly disparate yet well-known risk conditions, we can reduce PTB and the subsequent race/ethnic disparities.

ELIGIBILITY:
Inclusion Criteria:

* delivery of live born infant at <34 weeks of gestation in one of 18 Philadelphia area hospitals
* English or Spanish speaking
* Philadelphia residency
* not receiving operative sterilization before discharge from the hospital

Exclusion Criteria:

* N/A

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1136 (Actual)
Dates: Start 2004-11; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Reduction in PTB rate among women with a prior PTB can be achieved through interconceptional interventions targeting multiple as opposed to single risk factors. | Women in the intervention group will be assessed every 6 months through 24 months, unless they become pregnant, in which case they will be seen at 20 weeks EGA with their subsequent pregnancy.
  If women do not become pregnant during the evaluation period of 24 months, they will be seen for study visits every 6 months, and will be seen more often for intervention measures to take place, as needed. For those who become pregnant in the evaluation period, they will be assessed at 20 weeks EGA with their subsequent pregnancy, and asked to sign a release for their subsequent pregnancy records.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Culhane, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Webb DA, Mathew L, Culhane JF. Lessons learned from the Philadelphia Collaborative Preterm Prevention Project: the prevalence of risk factors and program participation rates among women in the intervention group. BMC Pregnancy Childbirth. 2014 Nov 1;14:368. doi: 10.1186/s12884-014-0368-0. PMID 25361563